CLINICAL TRIAL: NCT05504980
Title: The Effect of Repositioning Frequency Determined According to Body Mass Index on Pressure Ulcer Development Time: Randomized Controlled Trial
Brief Title: The Effect of Repositioning Frequency Determined According to BMI on Pressure Ulcer Development Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ebru Bulut, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AdnanMenderesU
Record Dates: First submitted 2022-08-03; First posted 2022-08-17 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Pressure Ulcer
Keywords: Nursing; Pressure ulcer; Body Mass Index; Reposition
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Patients in the intervention group will be given 30 degrees right lateral, supine, and 30 degrees left lateral positions, 1 hour apart, respectively.
  Interventions: Procedure: Repositioning
- Control group (No Intervention): Patients in the control group will be given 30 degrees right lateral, supine and 30 degrees left lateral positions, respectively, at 2 hour intervals according to the hospital routine practice.

INTERVENTIONS:
Procedure: Repositioning — Patients in the intervention group will be given 30 degrees right lateral, supine, and 30 degrees left lateral positions, 1 hour apart, respectively.
  Arms: İntervention group

SUMMARY:
The research will be carried out in an experimental/randomized controlled manner in order to determine the effect of the frequency of repositioning according to body mass index on the development of pressure ulcers in adults.

The sample size was determined as 66 people by power analysis. However, considering the losses, the number of patients included in the sample will 30% higher than the calculated value and it was planned to include 86 patients (43 intervention group, 43 control group) in the study. In the first 24 hours of hospitalization, body mass index will be calculated by skinfold thickness measurement, and data will be collected using the "Structured Questionnaire" for patients with no pressure sores, bedridden, high and very high risk according to the Braden Risk Assessment Scale. In calculating the body mass index of bedridden patients, skinfold thickness measurement, measurement of the interface pressure, which is the most important factor in the development of pressure sores, and calf circumference measurement will be performed to determine the decrease in muscle mass. The research will continue with position change applications between 08-24 hours every day of the week. Patients in the intervention group will be given 30 degrees right lateral, supine, and 30 degrees left lateral positions, 1 hour apart, respectively. Patients in the control group will be given 30 degrees right lateral, supine and 30 degrees left lateral positions, respectively, at 2 hour intervals according to the hospital routine practice. In the initial evaluation, the interface pressure will be measured with the Palm Q-Portable Interface Pressure Sensor from the occipital, scapula, sacrum, heels when the patients are in the supine position, and from the pressure points of the acromion, greater thoracantary, and malleolus prominence when they are in the 30 degrees right and 30 degrees left lateral positions. Patients will be evaluated first within the first 24 hours of hospitalization and on day 21 if a pressure ulcer develops or does not develop a pressure sore a second time.

If the study is successful, it is expected that pressure ulcers will not develop in patients who are positioned at more frequent intervals.

DETAILED DESCRIPTION:
Pressure sores usually occur with ischemia and cell death over bony prominences. It is one of the most common complications in bedridden patients in healthcare institutions worldwide. Its prevalence is used as a worldwide quality indicator and shows that pressure sores are a common health problem worldwide. Its incidence has been found in a wide range between 0% and 72.5% worldwide.

Pressure sores slow down the healing process, prolong the hospital stay, increase the risk of complications, and therefore adversely affect the quality of life of the patients. It increases the cost of maintenance and threatens life. Prevention of pressure sores and early diagnosis of possible tissue damage is important. For this, measures should be taken to eliminate or reduce the effects of risk factors by evaluating them correctly.

In the researches, the importance of body mass index, which plays a role in the development of pressure sores, has been determined. External pressure, which varies according to the body mass index, the physical characteristics of the patient and the characteristics of the support surface used, is the most important factor that plays a role in the development of pressure sores. Pressure sores occur due to external pressure.

The interface pressure, which occurs during the transmission of external pressure to the subcutaneous tissues between the support surface and the skin, may be different in people with different body structures. In studies, it is stated that collagen, muscle mass, adipose tissue density and body mass index around the capillaries affect the interface pressure. It is known that the density of collagen, muscle mass and adipose tissue is different in people with different body mass indexes.

It is important to keep the interface pressure low to allow the return of blood flow to prevent the formation of pressure-related wound.

For this, it is thought that by changing the frequency of repositioning, the interface pressure will prevent blood flow for a long time and tissue damage will be prevented.

ELIGIBILITY:
Inclusion Criteria:

* Bedridden (1 and 2 points from the activity and movement subheadings of the Braden Risk Assessment Scale)
* Pressure ulcer not yet developed
* In the first 24 hours of hospitalization, it was evaluated according to the Braden Risk Assessment Scale and determined to be at high risk (range of 10-12 points) for the development of pressure ulcers

Exclusion Criteria:

* With hip fracture
* The position is not considered appropriate by the physician.
* Connected to Mechanical Ventilator
* Presence of septic shock
* Albumin value ≤3.5 mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The rate of pressure ulcer development is changed in patients who are positioned more frequently. | 21 days
  If the study is successful, it is expected that the pressure ulcer development time will be prolonged or pressure ulcer will not develop in patients who are positioned more frequently.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Bulut, Researcher, Principal Investigator — Researcher; Zeynep Günes, Professor, Study Director — Researcher
Locations (1):
- Aydin Adnan Menderes University Research and Application Hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kimura N, Nakagami G, Minematsu T, Sanada H. Non-invasive detection of local tissue responses to predict pressure ulcer development in mouse models. J Tissue Viability. 2020 Feb;29(1):51-57. doi: 10.1016/j.jtv.2019.11.001. Epub 2019 Nov 4. PMID 31757582
- [Result] Kim S, Kim M, Lee Y, Kim B, Yoon TY, Won CW. Calf Circumference as a Simple Screening Marker for Diagnosing Sarcopenia in Older Korean Adults: the Korean Frailty and Aging Cohort Study (KFACS). J Korean Med Sci. 2018 Apr 26;33(20):e151. doi: 10.3346/jkms.2018.33.e151. eCollection 2018 May 14. PMID 29760608
- [Result] Mervis JS, Phillips TJ. Pressure ulcers: Pathophysiology, epidemiology, risk factors, and presentation. J Am Acad Dermatol. 2019 Oct;81(4):881-890. doi: 10.1016/j.jaad.2018.12.069. Epub 2019 Jan 18. PMID 30664905
- [Result] Mervis JS, Phillips TJ. Pressure ulcers: Prevention and management. J Am Acad Dermatol. 2019 Oct;81(4):893-902. doi: 10.1016/j.jaad.2018.12.068. Epub 2019 Jan 18. PMID 30664906
- [Result] Seo Y, Roh YS. Effects of pressure ulcer prevention training among nurses in long-term care hospitals. Nurse Educ Today. 2020 Jan;84:104225. doi: 10.1016/j.nedt.2019.104225. Epub 2019 Oct 23. PMID 31698290
- [Result] Saghaleini SH, Dehghan K, Shadvar K, Sanaie S, Mahmoodpoor A, Ostadi Z. Pressure Ulcer and Nutrition. Indian J Crit Care Med. 2018 Apr;22(4):283-289. doi: 10.4103/ijccm.IJCCM_277_17. PMID 29743767
- [Result] Neloska L, Damevska K, Nikolchev A, Pavleska L, Petreska-Zovic B, Kostov M. The Association between Malnutrition and Pressure Ulcers in Elderly in Long-Term Care Facility. Open Access Maced J Med Sci. 2016 Sep 15;4(3):423-427. doi: 10.3889/oamjms.2016.094. Epub 2016 Aug 22. PMID 27703567
- [Result] Hyun S, Li X, Vermillion B, Newton C, Fall M, Kaewprag P, Moffatt-Bruce S, Lenz ER. Body mass index and pressure ulcers: improved predictability of pressure ulcers in intensive care patients. Am J Crit Care. 2014 Nov;23(6):494-500; quiz 501. doi: 10.4037/ajcc2014535. PMID 25362673
- [Result] Coleman S, Nixon J, Keen J, Wilson L, McGinnis E, Dealey C, Stubbs N, Farrin A, Dowding D, Schols JM, Cuddigan J, Berlowitz D, Jude E, Vowden P, Schoonhoven L, Bader DL, Gefen A, Oomens CW, Nelson EA. A new pressure ulcer conceptual framework. J Adv Nurs. 2014 Oct;70(10):2222-34. doi: 10.1111/jan.12405. Epub 2014 Mar 31. PMID 24684197
- [Result] Bhattacharya S, Mishra RK. Pressure ulcers: Current understanding and newer modalities of treatment. Indian J Plast Surg. 2015 Jan-Apr;48(1):4-16. doi: 10.4103/0970-0358.155260. PMID 25991879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT05504980/Prot_SAP_001.pdf